CLINICAL TRIAL: NCT02976636
Title: Parent Training Program to Improve Outcomes in Childhood Obesity Treatment
Brief Title: Reinforced Enhanced - Families Responsibility Education Support and Health
Acronym: Re-FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kay Rhee, Associate Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DK106157 (NIH); R01DK106157 (NIH)
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Obesity
Keywords: Obesity treatment; Parenting training; Parenting style; Family-based behavioral therapy
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will not know which arm of the study each family is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-based behavioral therapy (FBT) (Active Comparator): Family-based behavioral therapy for pediatric weight loss
  Interventions: Behavioral: Family-based behavioral therapy
- Parenting training and FBT (Experimental): Family-based behavioral therapy for pediatric weight loss + parenting training to enhance outcomes
  Interventions: Behavioral: Family-based behavioral therapy; Behavioral: Parenting training

INTERVENTIONS:
Behavioral: Family-based behavioral therapy — Traditional family-based, group-based behavioral therapy for weight loss. Parent and child groups will be held separately. Intervention will consist of 20 sessions: 16 weekly sessions, and then every other week for 4 sessions.
  Other Names: FBT; FRESH
Behavioral: Parenting training — Parenting skills training for parents. Parent and child groups will be held separately and only parents will receive this training. Children will not receive any additional materials. Intervention will consist of 20 sessions: 16 weekly sessions, and then every other week for 4 sessions.
  Other Names: Re-FRESH; FBT + PT
  Arms: Parenting training and FBT

SUMMARY:
The purpose of this application is to evaluate whether a pediatric weight control program that incorporates comprehensive parenting training with behavioral therapy can increase weight loss in children compared to traditional family-based behavioral therapy programs. Since certain parenting styles are associated with greater weight loss during interventions and appear to enhance the impact of key behavioral strategies, adding parenting training to these interventions may increase the overall effectiveness of these programs and increase our ability to help children obtain a healthy weight. This project could result in identifying an improved method of pediatric obesity treatment that provides additional benefits to the growth and development of children via improved self-regulatory behaviors.

DETAILED DESCRIPTION:
Authoritative parenting style has been associated with decreased obesity risk in children, increased weight loss during interventions, and can modify the delivery and impact of weight control strategies, making them more effective. At this time, gold-standard treatment for childhood obesity is family-based behavioral therapy (FBT). This treatment relies on behavioral strategies and the use of praise and a positive reinforcement system to change eating and activity behaviors, but does not target other aspects of parenting. Broadening parenting instruction to include effective limit-setting behaviors, parent-child communication, and authoritative parenting may increase parents' confidence and ability to successfully make behavior changes and modify the impact of the behavioral strategies being used. In this application, the investigators propose to test the efficacy of a 20-week weight control program that combines traditional family-based behavioral therapy with comprehensive parenting training (FBT-PT) and compare it to traditional family-based behavioral therapy (FBT). The investigators hypothesize that there will be an additive effect of parenting training such that FBT-PT will have a greater effect on child weight loss (measured by BMI z-score) than traditional FBT. In addition, the investigators will measure parenting style, parenting strategies, behavioral strategies, and child factors (like impulsive behavior and temperament) to better understand the mediators and moderators of weight loss. These measures will be obtained by standard self-report measures and videotape encounters, allowing one to more objectively measure parenting dimensions. Clinical outcomes, like drop-out and acceptability, will also be assessed from the two treatment arms. The purpose of this study is to evaluate the effect of adding a comprehensive parenting training to traditional FBT. If successful, this program will be able to increase our ability to help children successfully lose weight.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 7 and 12 years old;
2. BMI ≥85th percentile but <100% overweight, so as to limit those children who are morbidly obese and are in need of more intense medical treatment;
3. Children with mothers who are willing to attend 20 weekly group sessions and be randomized to either treatment arm;
4. Have at least one parent who is overweight or obese (BMI≥25); and
5. Parents who speak English at a 5th grade level.

Exclusion Criteria:

1. Children with serious medical conditions that affect their weight;
2. Children taking medication that affect appetite or weight;
3. Children with severe developmental delay or disability that would affect participation;
4. Children or parents with psychological illness that would limit treatment participation;
5. Families who will move out of the area within the time frame of the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Change in BMI percentile | 6 months and 18 months
  Change in BMI percentile at the end of treatment and follow-up period

SECONDARY OUTCOMES:
Percent of families who Drop-out of study | 6 months
  Difference in percent of families who drop-out between groups
Child Report of Parent Behavior Inventory | 6 months and 18 months
  Change in parenting style from baseline to post-treatment and follow-up between groups
Percentage of sessions attended between groups | 6 months
  Difference in percentage of sessions attended between groups
Percent of families who adhered to treatment goals | 6 months
  Difference in percent of families who adhered to treatment goals between groups
Child feeding questionnaire | 6 months and 18 months
  Change in child feed behaviors from baseline to post-treatment and follow-up between groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rhee KE, Corbett T, Patel S, Eichen DM, Strong DR, Kang-Sim E, Anderson CAM, Marcus BH, Boutelle KN. Parenting Training Plus Behavioral Treatment for Children With Obesity: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e258398. doi: 10.1001/jamanetworkopen.2025.8398. PMID 40323600